CLINICAL TRIAL: NCT05708326
Title: Does Timing Matter? A Case Crossover Study of Intermittent Fasting in Patients With CLL/SLL at BC Cancer- Victoria
Brief Title: A Case Crossover Study of Intermittent Fasting in CLL/SLL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: BC Cancer Foundation (Other); University of Victoria (Other)
Responsible Party: Principal Investigator, Eleah Stringer, Dietitian Investigator, British Columbia Cancer Agency
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: H21-02145
Record Dates: First submitted 2022-12-21; First posted 2023-02-01 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Chronic Lymphocytic Leukemia (CLL); Small Lymphocytic Lymphoma (SLL)
Keywords: diet; nutrition; intermittent fasting; time restricted feeding; oncology; autophagy; metabolomics
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Intermittent Fasting; Neoplasms | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Participants will have previously completed the first arm (trial of the 16/8 intermittent fasting method), and are now invited to the second arm (the 5:2 Method), serving as their own control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5:2 Method (Experimental): Participants will follow the 5:2 Method (an intermittent fasting regimen) for a 90 day duration. This entails eating ad libitum for five days per week ("normal days") and limiting total calorie intake to 800kcals per day ("fasting days") for the remaining two days per week. The fasting days can be sequential or dispersed throughout the week, based on patient preference.
  Interventions: Behavioral: 5:2 Method (intermittent fasting regimen)
- 16/8 Method (Active Comparator): Participants will have already followed the 16/8 Method (an intermittent fasting regimen) for a minimum of six days per week for a 90 day duration. This entailed limiting the eating hours to an 8-hour window, then fasting for the remaining 16 hours per day, with the last time of intake being 8pm.
  Interventions: Behavioral: 16/8 Method (intermittent fast regimen)

INTERVENTIONS:
Behavioral: 5:2 Method (intermittent fasting regimen) — Participants will follow the 5:2 Method (an intermittent fasting regimen) for a 90 day duration. This entails eating ad libitum for five days per week ("normal days") and limiting total calorie intake to 800kcals per day ("fasting days") for the remaining two days per week. The fasting days can be sequential or dispersed throughout the week, based on patient preference.
  Arms: 5:2 Method
Behavioral: 16/8 Method (intermittent fast regimen) — Participants will have already followed the 16/8 Method (an intermittent fasting regimen) for a minimum of six days per week for a 90 day duration. This entailed limiting the eating hours to an 8-hour window, then fasting for the remaining 16 hours per day, with the last time of intake being 8pm.
  Arms: 16/8 Method

SUMMARY:
The purpose of this study is to compare the 16/8 intermittent fasting method with the 5:2 Method in a subset of patients with chronic lymphocytic leukemia or small lymphocytic lymphoma at BC Cancer- Victoria. The purpose is to find out which is the preferred method by patients and which has the greatest effect on:

* cancer cells (lymphyocyte count),
* metabolism (autophagy activation),
* inflammation (CRP),
* gut microbiome (metabolomic analysis).

Participants will have already completed our previous trial, "Intermittent Fasting in CLL/SLL" (ClinicalTrials.gov Identifier: NCT04626843) where they followed the 16/8 Fasting Method followed by a minimum of a 3 months washout period, and will now follow the 5:2 Method for 90 days. The same samples and outcome measures will be collected in order to directly compare the two diets in the same patient cohort.

DETAILED DESCRIPTION:
BACKGROUND: Interest in intermittent fasting (IF) is growing rapidly for its potential to improve health outcomes. IF is a diet regime that cycles between fasting and eating for a defined period. There are many variations of IF, most altering the length of the fasting window but some may include caloric restriction.

The investigators are nearing completion a feasibility study on the effects of IF on chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) at BC Cancer- Victoria. This clinical trial, "IF in CLL/SLL" (ClinicalTrials.gov Identifier: NCT04626843) investigates the biochemical effects of the 16/8 Method on CLL/SLL tumor control, markers of inflammation, and autophagy induction in a case-controlled study. Preliminary findings demonstrate excellent compliance and early feedback and findings are overwhelmingly positive. It is unknown, however, how the 16/8 Method compares to other IF regimens in terms of patient acceptability and biologic effects.

OBJECTIVE: The aim is to examine the two most common regimens, the 16/8 Method (16 hr fast) and the 5:2 Method (2 day per week of caloric restriction of 800 kcals). The primary research questions are, which IF strategy has the greatest effect on, (1) tumour burden (lymphocyte count), (2) autophagy induction and gut microbiome composition, (3) inflammation, (4) and is preferred by patients.

METHODS: This study is an extension of the investigators' current, single-arm trial to expand to a case crossover design, allowing each participant to serve as their own control. Following completion of a 90 day trial on the 16/8 Method during the "Intermittent Fasting in CLL/SLL" study (ClinicalTrials.gov Identifier: NCT04626843) and following a minimum of a 3 month washout period, participants will now follow the 5:2 Method for 90 days. Data collection will match previous current study protocol to allow for statistical comparison between lymphocyte count, inflammation, metabolomic profiles, autophagy status, and the gut microbiome (optional). Participants will complete a semi-structured interview on their experiences with the 16/8 Method and 5:2 Method that will be qualitatively analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL or SLL
* Age < 85 years
* Peripheral blood lymphocytes >20 x 109/L
* Hemoglobin > 90g/L
* Platelets > 90 x 10*9/L
* BMI of >=20kg/m2
* ECOG Performance Status >=2
* Completion of "IF in CLL/SLL Study" (ClinicalTrials.gov Identifier: NCT04626843) followed by minimum of 3 month ad libitum eating

Exclusion Criteria:

* Patient unable to give consent
* Patient on medications required to be taken with food during the fasting window
* Pregnancy
* Diabetes mellitus
* BMI drop to < 18.5kg/m2 at any time during study
* Anti-lymphoma therapy within the past 3 months
* Expected to require initiation of anti-lymphoma therapy within the next 3 months

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in lymphocyte count [ Time Frame: Within 3 months pre-intervention, monthly during intervention, 1 month post-intervention ] | Within 3 months pre-intervention, monthly during intervention, 1 month post-intervention
  Changes in lymphocyte count will be measured between each peripheral blood draw and also compared to the former results as part of the "IF in CLL/SLL Study" (ClinicalTrials.gov Identifier: NCT04626843).
Change in inflammation | Within 3 months pre-intervention, monthly during intervention, 1 month post-intervention
  Changes in c-reactive protein (CRP) will be measured between each peripheral blood draw and also compared to the former results as part of the "IF in CLL/SLL Study" (ClinicalTrials.gov Identifier: NCT04626843).
Change in metabolomic profiles (optional) | Day 1 (start/baseline) and day 90 (end/final) of intervention
  Changes in abundance of stool metabolites will be measured between each stool sample and between the two interventional arms. This includes, but is not limited to, an established short-chain fatty acid and bile acid panel that analyzes 77 and 10 unique metabolites, respectively.
Change in autophagy status | Time Frame: Within 3 months pre-intervention, monthly during intervention, 1 month post-intervention
  This includes standard flow cytometric analysis of lymphocyte subsets: a panel established by the Human Immunology Consortium Project as well as additional in-house markers to enumerate the frequency of lymphocytes before and at various time points post-treatment. The extent of autophagy will be tested by performing cytometry and western blotting assays using LC3II and p62 as readouts. Total cell counts in different lymphocyte subsets including, but not limited to, cluster of differentiation (CD) 3, CD8, CD4, CD20, CD19, and forkhead box P3 (FoxP3) will be assayed in conjugation with glucose uptake and mitochondrial function.
Changes in immune cell gene expression profiles | Time Frame: Within 3 months pre-intervention, monthly during intervention, 1 month post-intervention
  Changes in expression profiles of selected immune cell genes

SECONDARY OUTCOMES:
Change in gut microbiome (optional) | Day 1 (start/baseline) and day 90 (end/final) of intervention
  Stool samples to identify baseline and fasting-induced changes in abundance and repertoire of the gut microbiota.

CONTACTS AND LOCATIONS:
Overall Officials: Nicol Macpherson, MD, PhD, FRCPC, Principal Investigator — BC Cancer and University of British Columbia
Locations (1):
- Eleah Stringer, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stringer E, Lum JJ, Macpherson N. Intermittent Fasting in Cancer: a Role in Survivorship? Curr Nutr Rep. 2022 Sep;11(3):500-507. doi: 10.1007/s13668-022-00425-0. Epub 2022 May 31. PMID 35639262